CLINICAL TRIAL: NCT01325103
Title: Phase 1 Study of Autologous Bone Marrow Stem Cell Transplantation in Patients With Spinal Cord Injury
Brief Title: Autologous Bone Marrow Stem Cell Transplantation in Patients With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sao Rafael (Other)
Collaborators: Oswaldo Cruz Foundation (Other); Irep Sociedade de Ensino Superior Médio e Fundamental Limitada (Other); Hospital Espanhol (Network)
Responsible Party: Principal Investigator, Ricardo Ribeiro dos Santos, Phase 1 Study of Autologous Bone Marrow Stem Cell Transplantation in Patients With Spinal Cord Injury, Hospital Sao Rafael
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCI-001
Record Dates: First submitted 2011-03-28; First posted 2011-03-29 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2014-05

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord injury; Mesenchymal stem cells; Bone marrow
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Stem Cell Transplantation

STUDY DESIGN:
Intervention Model Description: Mesenchymal stem cell transplantation.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cell Transplantation (Experimental): Patients with spinal cord injury that will undergo autologous bone marrow stem cell transplantation.
  Interventions: Procedure: Stem Cell Transplantation

INTERVENTIONS:
Procedure: Stem Cell Transplantation — All patients will undergo autologous bone marrow stem cell transplantation into the lesion area.
  Other Names: BMMSC - Bone Marrow Mesenchymal Stem Cells.

SUMMARY:
This research investigates the use of autologous bone marrow stem cells in patients with spinal cord injury.

DETAILED DESCRIPTION:
The aim of this study is to evaluate autologous bone marrow stem cells transplantation as a safe and potentially beneficial treatment for patients with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years old
* Traumatic spinal cord injury at the thoracic or lumbar level
* Classification Frankel A
* Indication for spinal surgery for traumatic lesions of bone

Exclusion Criteria:

* Section of the spinal anatomy
* Open injuries
* Active infectious diseases
* Terminal patients
* Neurodegenerative diseases
* Primary hematologic diseases
* Bone reflecting increased risk for spinal puncture
* Coagulopathies
* Hepatic dysfunction
* Pregnancy
* Other medical complications that contraindicate surgery, including major respiratory complications
* Participation in another clinical trial
* Use of metal implants close to vascular structures (such as cardiac pacemaker or prosthesis) that contraindicate MRI

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Feasibility and safety of bone marrow stem cell transplantation in patients with spinal cord injury | Six months

SECONDARY OUTCOMES:
Functional improvement in muscle strength | Six months
  Functional improvement in muscle strength assessed by the Frankel scale.
Improvement of sphincters control. | Six months
  Improvement of sphincters control (anal and bladder).

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo R. dos Santos, MD, PhD, Principal Investigator — Hospital Sao Rafael; Milena Botelho P. Soares, PhD, Study Director — Hospital Sao Rafael; Marcus Vinícius P. Mendonça, MD, Study Chair — Hospital Sao Rafael; Cláudia B. Pinheiro, PhD, Study Chair — Hospital Sao Rafael; Ticiana X. Ferreira, MD, Study Chair — Hospital Sao Rafael; Cristiane F. Villarreal, PhD, Study Chair — Hospital Sao Rafael; Luiz Flávio M. Silva, MD, Study Chair — Hospital Sao Rafael; Marco A. Almeida, MD, Study Chair — Hospital Sao Rafael; Ubirajara B. Júnior, MD, PhD, Study Chair — Hospital Sao Rafael
Locations (1):
- Hospital São Rafael, Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Derived] Mendonca MV, Larocca TF, de Freitas Souza BS, Villarreal CF, Silva LF, Matos AC, Novaes MA, Bahia CM, de Oliveira Melo Martinez AC, Kaneto CM, Furtado SB, Sampaio GP, Soares MB, dos Santos RR. Safety and neurological assessments after autologous transplantation of bone marrow mesenchymal stem cells in subjects with chronic spinal cord injury. Stem Cell Res Ther. 2014 Nov 17;5(6):126. doi: 10.1186/scrt516. PMID 25406723